CLINICAL TRIAL: NCT06078956
Title: ABL90 FLEX PLUS Method Comparison Study for pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb in Whole Blood in Adult Population.
Brief Title: ABL90 Flex Plus Method Comparison Study_Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DC-083659
Record Dates: First submitted 2023-02-14; First posted 2023-10-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Diagnostic Test
Keywords: Blood gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigational Device (Active Comparator)
  Interventions: Device: Measuring of analytes
- Predicate device (Other)
  Interventions: Device: Measuring of analytes

INTERVENTIONS:
Device: Measuring of analytes — Method Comparison Study for pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb in whole blood in adult population.

SUMMARY:
The goal of this clinical trial is to validate performance claims for method comparison for the ABL90 FLEX PLUS for pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb in heparinized whole blood in a Point of Care (POC) setting.

DETAILED DESCRIPTION:
The main question it aims to answer is:

To quantify the relationship using comparison measurement from the same sample between ABL90 FLEX PLUS and the predicate device within the reportable range for all 15 parameters in heparinized arterial and venous patient whole blood in syringe measuring mode (S65, SP65) and heparinized capillary whole blood samples in capillary measuring mode (C65).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years or older.
* Informed consent collected from subject or from relative(s) able to understand information given and willing and able to voluntary give their consent to participate in this study.
* The subject will provide blood samples from the existing Aand/ or V-lines, and/or from a finger stick.
* Subject evaluated as suitable according to the protocol to enroll in the study by principal investigator or designee.

Exclusion Criteria:

* Subject where sample collection is evaluated by principal investigator or designee to impose an unnecessary risk.
* Subject, who is pregnant or breastfeeding.
* Subject, who has an invalid written informed consent or has withdrawn consent.
* Subject who has already provided successful measurements of arterial, venous and capillary samples, to cover both syringe modes and the capillary mode
* Subjects taking medications listed in Appendix 1 with last dose within 72 hours, should be excluded due to interference.
* Subjects with known infectious disease such as Hepatitis C and HIV (in order to ensure the operator safety).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Slope, R^2 and bias at medical decision points | 6-9 months
  Primary Endpoints: Slope, R^2 and bias at medical decision points for each combination of modes and sample type, across sites

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Bærentzen, PhD, Study Director — Radiometer Medical ApS
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No